CLINICAL TRIAL: NCT01146457
Title: The Optimal Dosage of Intrathecal Morphine for Peripartum Analgesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Hess, Chief of Obstetric Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009P000197
Record Dates: First submitted 2010-06-14; First posted 2010-06-17 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Labor Pain
Keywords: Obstetric anesthesia; labor analgesia; morphine; epidural analgesia
MeSH Terms: conditions — Labor Pain | interventions — Morphine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline
- Morphine 25 (Active Comparator)
  Interventions: Drug: Morphine
- Morphine 50 (Active Comparator)
  Interventions: Drug: Morphine
- Morphine 75 (Active Comparator)
  Interventions: Drug: Morphine
- Morphine 100 (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Active dosage
  Other Names: Dose of morphine added to solution
  Arms: Morphine 100; Morphine 25; Morphine 50; Morphine 75
Drug: Saline — Saline Control
  Other Names: Saline added to solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the ideal dosage of intrathecal morphine for intra and post partum analgesia, while minimizing the side effect profile.

DETAILED DESCRIPTION:
Regional anesthesia techniques such as combined spinal epidural (CSE) analgesia are very effective for the management of intrapartum pain. The advantages of these techniques are that they are safe when properly conducted and that they provide excellent analgesia while allowing the patient to remain awake and participate in the labor and delivery. The risks of maternal aspiration and fetal drug depression associated with general anesthesia are minimized. Finally, the effective analgesia associated with regional techniques blunt the hemodynamic effects caused by painful contractions and reduce maternal catecholamines, resulting in increased placental perfusion.1

Opioids in combination with local anesthetics in the spinal space provide effective pain relief during labor with minimal side effects. The advantages of spinal opioid administration include lack of motor blockade and faster onset of analgesia.2 In addition, since the opiate receptors are in the spinal space, a smaller amount of opioid can be used to provide excellent pain relief while minimizing the side effects. At Beth Israel Deaconess Medical Center (BIDMC), the obstetric anesthesiology group uses a standard spinal dosing for CSE during labor which includes: 1 ml of 0.25% bupivicaine with 12.5 mcg of fentanyl.

Yeh and colleagues have found that morphine 150 mcg added to the fentanyl-bupivicaine spinal injection can prolong the duration of spinal analgesia but was associated with increased side effects. 3 The side effect profile of spinal narcotics include: nausea, vomiting, pruritus, and urinary retention. Although these side effects for the most part can be easily treated, they can be bothersome to the post partum patient. In a previous study performed from our institution, the addition of 100 mcg of morphine to spinal bupivicaine and fentanyl reduced the rate of breakthrough pain during labor analgesia and prolonged the time to first request for supplementation. Overall, it was found that the incidence of side effects was low but the group that received the spinal morphine did have more nausea and vomiting compared with the placebo group. 4

In this current investigation, we would like to assess whether an even smaller dose of spinal morphine would provide an effective, pain free recovery from vaginal delivery while decreasing the incidence of side effects, specifically nausea and vomiting. We would like to perform a formal dose response study to identify the ideal dose of intrathecal morphine that would not compromise the pain relief during labor while minimizing the side effects.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy,
* at least 36 weeks gestational age,
* active labor (≤ 5 cm dilation) requesting neuraxial analgesia,
* ASA I or II,
* not currently taking pain medications.

Exclusion Criteria:

* multiple gestation,
* preterm labor,
* systemic opioids in the past 4 hours,
* chronic pain syndromes,
* chronic opioid use,
* contraindications to regional anesthesia,
* allergies to opioids,
* significant co existing medical problems,
* severe pregnancy induced hypertension,
* sedatives,
* magnesium therapy,
* diabetes type 1.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2010-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Hess, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine 25: Morphine 25 micrograms: Active dosage
- Morphine 50: Morphine 50 micrograms: Active dosage
- Morphine 75: Morphine 75 micrograms: Active dosage
- Morphine 100: Morphine 100 micrograms: Active dosage
Period: Overall Study
Arm/Group | Placebo | Morphine 25 | Morphine 50 | Morphine 75 | Morphine 100
Started | 19 | 17 | 21 | 13 | 13
Completed | 19 | 17 | 20 | 13 | 13
Not Completed | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Saline control
- Morphine 25: Morphine 25 micrograms
- Morphine 50: Morphine 50 micrograms
- Hine 75: Morphine 75 micrograms
- Morphine 100: Morphine 100 micrograms
- Total: Total of all reporting groups
Arm/Group | Placebo | Morphine 25 | Morphine 50 | Hine 75 | Morphine 100 | Total
Number analyzed (Participants) | 19 | 17 | 21 | 13 | 13 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (5.3) | 31.5 (5.3) | 31.3 (6.6) | 32.5 (5.5) | 32.4 (5.7) | 32.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 21 | 13 | 13 | 83
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Breakthrough Pain
Description: Rate of breakthrough pain is the number of episodes of breakthrough pain divided by the number of hours of labor. Time measured from placement of the neuraxial anesthetic, until delivery of the neonate. Because duration of labor is different for all patients, the rate of breakthrough pain per hour is used as the primary outcome.
Time Frame: Participants were followed for the duration of delivery, an average of 7 hours
Measure: Mean (Standard Deviation); unit: episodes of breakthrough pain per hour
Groups:
- Control: Saline Control
- Morphine 75: Morphine 75 micrograms
Arm/Group | Control | Morphine 25 | Morphine 50 | Morphine 75 | Morphine 100
Number analyzed (Participants) | 19 | 17 | 21 | 13 | 13
episodes of breakthrough pain per hour | 0.25 (0.29) | 0.28 (0.35) | 0.25 (0.25) | 0.23 (0.26) | 0.17 (0.21)

ADVERSE EVENTS:
Arm/Group | Placebo | Morphine 25 | Morphine 50 | Morphine 75 | Morphine 100
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17 | 0/21 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17 | 0/21 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No